CLINICAL TRIAL: NCT03380611
Title: Effects of Wakame and Spirulina Consumption on Intestinal Cholesterol Absorption in Non- Hypercholesterolemic Men and Women
Brief Title: Algae and Cholesterol Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: METC 17-3-022
Record Dates: First submitted 2017-12-07; First posted 2017-12-21 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2017-12

CONDITIONS: Intestinal Cholesterol Absorption

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wakame (Experimental): Subjects will receive capsules containing wakame
  Interventions: Dietary Supplement: Wakame
- Spirulina (Experimental): Subjects will receive capsules containing spirulina
  Interventions: Dietary Supplement: Spirulina
- Control (Placebo Comparator): Subjects will receive capsules containing microcrystalline cellulose
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Wakame — Consumption of 4.8 grams wakame per day for 17 days
  Other Names: Undaria pinnatifida
  Arms: Wakame
Dietary Supplement: Spirulina — Consumption of 4.8 grams spirulina per day for 17 days
  Other Names: Arthrospira
  Arms: Spirulina
Dietary Supplement: Control — Consumption of microcrystalline cellulose for 17 days
  Arms: Control

SUMMARY:
The primary objective of this study is to investigate the effects of wakame and spirulina consumption on intestinal cholesterol absorption.

DETAILED DESCRIPTION:
Objectives:

Secondary objectives are to investigate the effects of wakame and spirulina consumption on fasting markers for lipid metabolism, glucose metabolism and blood pressure.

Study design:

This study is a double-blinded, randomized, placebo-controlled, crossover intervention trial consisting of three intervention periods of 17 days each, separated by a minimum washout period of 14 days.

Study population:

The study population will consist of 37 healthy, non-hypercholesterolemic men and women aged between 18 and 70 years.

Intervention:

All subjects will receive wakame, spirulina and placebo capsules in randomized order. Subjects will be asked to consume 12 capsules per day for 17 days, which is equal to 4.8 grams of wakame or spirulina a day.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years;
* BMI between 18 and 30 kg/m2;
* Non-smoking;
* No elevated serum triacylglycerol concentrations (< 4.5 mmol/L);
* Willing to comply to the study protocol during the study;
* Agreeing to be informed about medically relevant personal test-results.

Exclusion Criteria:

* Not willing to abstain from any algae and/or seaweed consumption or algae/seaweed containing products two weeks before the start and during the trial;
* Use of plant-sterol/stanol-enriched foods (e.g. Becel Proactive) or supplements in the four weeks prior to the screening and/or during the study;
* Use of cholesterol or lipid-lowering medications (e.g. statins, bile-acid sequestrates, cholesterol absorption inhibitors);
* Use of any kind of medication or a medically prescribed diet, which can interfere with the study;
* Use of oral antibiotics in 40 days or less prior to the start of the study;
* Use of food supplements that might interfere with study measurements (judged by the principal investigator) in four weeks or less prior to the start of the study;
* Indications of treatment according to the Standard for Cardiovascular Risk Management from the Dutch General Practitioners community;
* Any medical condition that might interfere with study (measurements), judged by the principal investigator, including cardiovascular diseases or events (e.g. acute myocardial infarction or cerebro-vascular accident), diabetes, asthma, COPD, rheumatoid arthritis, and gastro-intestinal diseases (e.g. inflammatory bowel disease);
* Unstable body weight (weight gain or loss > 3 kg in the past 3 months);
* Females who are pregnant, breast feeding or who may wish to become pregnant during the study;
* Consumption of > 14 (males) or > 10 (females) alcoholic consumptions a week;
* Reported intense sporting activities > 10 hours a week;

  ￼• Abuse of drugs;
* Participation in any other biomedical trial four weeks prior to the screening visit;
* Having donated >150 ml blood within 1 month prior to the screening visit, planning to donate blood during the study or within one month after finishing the study;
* Impossible or difficult to puncture as evidenced during the screening visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
Markers for intestinal cholesterol absorption | Difference in outcomes between interventions and control at 17 days
  Serum cholesterol-standardized campesterol concentrations will be measured as a marker for intestinal cholesterol absorption

SECONDARY OUTCOMES:
Lipids | Difference in outcomes between interventions and control at 17 days
  Several markers for fasting lipid metabolism, including total cholesterol, LDL cholesterol and HDL cholesterol, will be measured in blood samples
Markers for cholesterol synthesis | Difference in outcomes between interventions and control at 17 days
  Serum cholesterol-standardized lathosterol and desmosterol concentrations will be measured as a markers for cholesterol synthesis
Glucose concentrations | Difference in outcomes between interventions and control at 17 days
  Fasting plasma glucose concentrations will be determined
Blood pressure | Difference in outcomes between interventions and control at 17 days
  Systolic and diastolic blood pressure will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Mensink, Professor, Principal Investigator — Maastricht University Medical Center; Jogchum Plat, Professor, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands